CLINICAL TRIAL: NCT02518776
Title: Influence of Emotional Disorders and Executive on the Components Retrograde and Anterograde Episodic Memory in MS
Acronym: ITEMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09-016
Record Dates: First submitted 2015-08-06; First posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neuropsychological tests (Other)
  Interventions: Behavioral: Neuropsychological tests

INTERVENTIONS:
Behavioral: Neuropsychological tests — Neuropsychological tests

SUMMARY:
Multiple sclerosis (MS) is an inflammatory disease of the central nervous system responsible for physical disability but can also cause cognitive disturbances annoying social and professional life of patients with the disease. Various studies have shown that there was a breach of episodic memory, working memory, attention and executive functions regardless of the form of disease, disability or duration of disease progression.

The main objective of this study is to investigate the influence of emotional components and executive processes on the components retrograde and anterograde episodic memory (thanks to an original paradigm based on the emotional valence of the memory) in MS patients

ELIGIBILITY:
Inclusion Criteria:

* Men and women 30-60 years of age
* Definite MS (McDonald criteria revised in 2005)
* EDSS <6
* Sick Shapes: Relapsing multiple sclerosis, Primary progressive multiple sclerosis
* All durations evolution
* French Mother tongue
* Signature of informed consent

Exclusion Criteria:

* Other neurological conditions, previous psychiatric or developmental diagnosis of MS
* Head injury sequelae
* Chronic alcohol or drugs Taking
* EDSS greater than or equal to 6
* Secondary Progressive Form
* Push and / or treatment with corticosteroids within one month
* Treatments Amantadine, Modafinil introduced for less than 3 months
* Patient Trust
* Cognitive Assessment of less than one year (including in particular all or part of the balance sheet proposed in this project)
* Any visual motor deficit or incompatible with the award of cognitive tests
* For women, pregnancy, breastfeeding and / or lack of contraception (a pregnancy test will be done before the PET scan)
* Patient with indications against MRI

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-06; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
anterograde episodic memory: 3 scores of emotional ESR | baseline
  3 scores of emotional ESR
retrograde episodic memory: 9 scores TEMP emotional | baseline
  9 scores TEMP emotional

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurologie, Caen Hospital University, Caen, Basse-Normandie, France